CLINICAL TRIAL: NCT06960200
Title: Phototherapy for Non-responders to Oral Appliance Therapy for Obstructive Sleep Apnea
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00125341
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- NL C3 (Experimental)
  Interventions: Device: Phototherapy
- QN (Experimental)
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — Non-surgical laser therapy (phototherapy)
  Arms: NL C3; QN

SUMMARY:
Obstructive sleep apnea (OSA) is a medical condition where a person has great difficulty with breathing, or stops breathing all together, while asleep. This is a medical condition for which one of the current standard treatments is the use of a custom made dental appliance to help hold the person's airway open while asleep so that the person does not suffocate while sleeping. However, while the majority of OSA patients are able to tolerate the use of oral appliance therapy (OAT) for OSA, some patients are incomplete responders to OAT. These patients, despite having improvement, may still have a disease index above the diagnostic threshold for OSA.

Phototherapy (laser therapy) has been used as a method to stiffen the soft palate and parts of the tongue to prevent their collapse. This is a type of cold laser therapy that does not cut/ablate tissue (similar to healing laser therapies). This has been shown to help with both snoring and can also help with OSA, as soft palate and tongue collapse are common areas for where OSA occurs inside the airway. A recent pilot study has shown that phototherapy on its own may be able to treat selected patients with mild, moderate, or severe OSA. To our knowledge, there are no contraindications to combining phototherapy and dental sleep appliance therapy.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether phototherapy (nightlase/quiet night laser protocol) can change oral appliance therapy (OAT) incomplete responders into complete responders for the treatment of obstructive sleep apnea (OSA). Patients who are incomplete responders to OAT will become complete responders (as defined as a reduction of 50% and below 10) with the adjunctive use of phototherapy for OSA. Per the American Academy of Sleep Medicine, first line treatment for OSA is CPAP. Patients who are unable to tolerate CPAP or otherwise decline CPAP may be treated through OAT. However, which compliance with OAT is significantly greater than CPAP, overall efficacy of OAT is not as high as CPAP. Further treatment options for patients with are incomplete responders to OAT are limited (other options include surgical interventions such as bariatric surgery and/or jaw surgery). The use of phototherapy for OAT incomplete responders offers the possibility of changing the response pattern for these patients into complete response which may provide more complete treatment rather than partial management for their OSA. Data to be collected for this study will be standard data collected for dental sleep appliance therapy. This includes mandibular position (in digital impression form and as OJ and OB recordings), range of motion, side effects/adverse reactions, titrations (% and number), total time required for treatment, medical history, CBCT imaging, biographical data, phototherapy exposure settings, etc.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with OSA
* incomplete treatment with OAT/MAD

Exclusion Criteria:

* not diagnosed with OSA
* using CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
OSA disease index | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta T6G 2E1, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: No